CLINICAL TRIAL: NCT00940953
Title: A Randomized, Double-Blind, Placebo-Controlled, 3-Way Cross-Over Study Comparing Relative Efficacy of CE Budesonide+Azelastine & Rhinocort Aqua+Astelin Nasal Sprays Against Placebo in the Treatment of AR in an EEC Model
Brief Title: Compare Captisol-Enabled (CE) Budesonide + Azelastine Nasal Solution and Rhinocort Aqua + Astelin in an Environmental Exposure Chamber (EEC) Study of Allergic Rhinitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ligand Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: CDX313CT001; P2DS07001
Record Dates: First submitted 2009-07-15; First posted 2009-07-17 (Estimated); Last update posted 2012-10-04 (Estimated); Status verified 2012-10

CONDITIONS: Seasonal Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal | interventions — Budesonide; azelastine; SBE4-beta-cyclodextrin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Captisol-Enabled Budesonide + Azelastine (Experimental)
  Interventions: Drug: Budesonide + Azelastine
- Rhinocort Aqua+Astelin (Active Comparator)
  Interventions: Drug: Budesonide + Azelastine
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Budesonide + Azelastine — nasal spray, one spray per nostril at time 0 plus one spray Placebo
  Other Names: CDX-313; Captisol
  Arms: Captisol-Enabled Budesonide + Azelastine
Drug: Budesonide + Azelastine — nasal spray, one spray of each per nostril at time 0
  Other Names: Rhinocort Aqua; Astelin
  Arms: Rhinocort Aqua+Astelin
Drug: Placebo — nasal spray, one spray per nostril from each of 2 bottles at time 0
  Other Names: phosphate buffered saline solution
  Arms: Placebo

SUMMARY:
The primary objective of this study was to compare Placebo to Captisol-Enabled Budesonide + Azelastine in a single spray and two separate sprays (Budesonide + Azelastine) in patients with Seasonal Allergic Rhinitis exposed to controlled ragweed pollen.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a clinical history of SAR
* Adults (males and females) aged 18 to 65
* Patients must have documentation of a positive skin test within 12 months of screening to ragweed allergen defined by a positive case history and a positive skin prick and/or intradermal test for ragweed allergen.
* Non-pregnant, non-lactating females, or women who are post-menopausal or are naturally or surgically sterile
* Females of childbearing potential must have a confirmed absence of pregnancy according to a negative urine pregnancy test and must be using acceptable birth control methods
* In generally good health on the basis of medical history and physical examination.
* Willingness to attend all study visits.
* Capable of following and understanding instructions.
* Willing and able to provide written informed consent prior to initiation of any study procedures, including initiation of washout of any concomitant medications

Exclusion Criteria:

* Pregnancy, nursing, or plans to become pregnant or donate gametes (ova or sperm) for in-vitro fertilization
* Have clinically significant physical findings of nasal anatomical deformities causing greater than 50% obstruction based on the clinical estimate of the investigator, including nasal polyps, septal defects or other clinically significant respiratory tract malformations, recent nasal biopsy, nasal trauma, or surgery and atrophic rhinitis or rhinitis medicamentosa
* Previous participation in a budesonide study within 1 month prior to the Screening Visit.
* Currently participating in a clinical trial or has been exposed to an investigational treatment within the 30 days prior to the Screening Visit.
* A known hypersensitivity to any corticosteroid or any of the excipients in the formulation of the investigational drug (e.g., any adverse experience with budesonide, azelastine or the Captisol-containing products Vfend IV or Geodon IM).
* History of severe respiratory infection or disorder
* History of alcohol or drug abuse
* History of a positive test for HIV, hepatitis B or hepatitis C.
* Use of any of the prohibited medications within the identified exclusion periods
* Use of antibiotic therapy for acute conditions
* Initiation of immunotherapy or dose escalation during the study period.
* Non-vaccinated exposure to or active infection with chickenpox or measles within the 21 days preceding the Screening Visit.
* Exposure to systemic corticosteroids
* Use of topical corticosteroids in concentrations in excess of 1% hydrocortisone or equivalent
* History of epilepsy or seizures
* History of coronary heart disease, uncontrolled hypertension, or other clinically significant cardiovascular disease.
* Have any of the following conditions that are judged by the investigator to be clinically significant and/or affect the patient's ability to participate in the clinical trial:

  * Impaired hepatic function including alcohol related liver disease or cirrhosis
  * History of ocular disturbances (e.g., glaucoma or posterior subcapsular cataracts)
  * Any systemic infection
  * Hematological, renal, endocrine (except for controlled diabetes mellitis or postmenopausal symptoms or hypothyroidism)
  * Gastrointestinal disease
  * Malignancy (excluding basal cell carcinoma)
  * A current neuropsychiatric condition with or without drug therapy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2008-02; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Patient-rated Total Nasal Symptom Score | 10 mins, 20 mins, 30 mins, 40 mins, 60 mins, 90 mins, 120 mins and then every hour up to 10 hours post dose

SECONDARY OUTCOMES:
Patient-rated Total Symptom Score | 10 mins, 20 mins, 30 mins, 40 mins, 60 mins, 90 mins, 120 mins and then every hour up to 10 hours post dose
Patient-rated EEC-RQLQ assessment | -0.75 hours, 2 hours, 6 hours and 10 hours post dose

CONTACTS AND LOCATIONS:
Overall Officials: Deepen Patel, MD, Principal Investigator — Allied Research International - Cetero Research
Locations (1):
- Allied Research International - Cetero Research, Mississauga, Ontario, Canada